CLINICAL TRIAL: NCT01108250
Title: LOC387715/HTRA1 Variants in Polypoidal Choroidal Vasculopathy in a Korean Population
Acronym: PCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, clinical professor, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LOC387715/HTRA1
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Genotype

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polypoidal choroidal vasculopathy (Experimental): patients with polypoidal choroidal vasculopathy
  Interventions: Genetic: LOC387715/HTRA1 genotyping
- control (Active Comparator): control group with no polypoidal choroidal vasculopathy
  Interventions: Genetic: LOC387715/HTRA1 genotyping

INTERVENTIONS:
Genetic: LOC387715/HTRA1 genotyping — Genomic DNA was extracted from whole blood by standard methods. Genotyping was performed using SNP Genotyping Assays.
  Other Names: genotyping

SUMMARY:
This study is to investigate whether variants in the LOC387715 locus and the HtrA serine peptidase 1 (HTRA1) gene within the 10q26 locus are associated with polypoidal choroidal vasculopathy and whether they are associated with clinical patterns including angiographic phenotype in a Korean population.

DETAILED DESCRIPTION:
This is a cross-sectional case-control study. One hundred Korean patients with polypoidal choroidal vasculopathy and 100 control subjects were genotyped for the LOC387715 (rs10490924) and the HTRA1 gene polymorphism (rs11200638)

ELIGIBILITY:
Polypoidal choroidal vasculopathy group

Inclusion Criteria:

* patients older than 60 years of age at onset
* polyp-like terminal aneurysmal dilations with or without branching vascular networks in indocyanine green angiography and subretinal reddish-orange protrusions corresponding to polyp-like lesions

Exclusion Criteria:

* eyes with pathologic myopia, angioid streaks, central serous chorioretinopathy, and other retinal or choroidal diseases

Control group

Inclusion Criteria:

* individuals without retinal diseases and without any signs of polypoidal choroidal vasculopathy or age-related macular degeneration on the bases of comprehensive ophthalmic examination results

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Genotyping of LOC387715/HTRA1 of PCV and control groups | 4weeks
  to investigate whether variants in the LOC387715 locus and the HtrA serine peptidase 1 (HTRA1) gene within the 10q26 locus are associated with polypoidal choroidal vasculopathy (PCV)

SECONDARY OUTCOMES:
Indocyanine angiographic findings of polypoidal choroidal vasculopathy | 20 minutes
  The association of the risk allele of the LOC387715/HTRA1 and indocyanine angiographic characteristics of polypoidal choroidal vasculopathy including subretinal hemorrhage, pigment epithelial detachment, and serous retinal detachment.
Visual acuity using Snellen chart | 2 x 5 minutes
  To evaluate the association between visual acuity and genotype of polypoidal choroidal vasculopathy

CONTACTS AND LOCATIONS:
Overall Officials: In Taek Kim, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- In Taek Kim, Daegu, Kyungsangpookdo, South Korea

REFERENCES:
- [Background] Gotoh N, Nakanishi H, Hayashi H, Yamada R, Otani A, Tsujikawa A, Yamashiro K, Tamura H, Saito M, Saito K, Iida T, Matsuda F, Yoshimura N. ARMS2 (LOC387715) variants in Japanese patients with exudative age-related macular degeneration and polypoidal choroidal vasculopathy. Am J Ophthalmol. 2009 Jun;147(6):1037-41, 1041.e1-2. doi: 10.1016/j.ajo.2008.12.036. Epub 2009 Mar 9. PMID 19268887
- See also: genetics home reference — http://ghr.nlm.nih.gov/
- See also: MedlinePlus related topics — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v:project=medlineplus&query=loc387715